CLINICAL TRIAL: NCT02894801
Title: Multistate Relative Survival Modeling of Colorectal Cancer Progression and Mortality
Brief Title: Multistate Relative Survival Model
Acronym: MRS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PIOC 2015
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Colorectal cancer (CRC) has high incidence and is associated with high case fatality. In France, the 5-year survival, pooled across all cancer stages at diagnosis, ranges from 57% in men to 60% in women. About one third of patients diagnosed with CRC will develop a metachronous recurrence during the following years. It is of paramount importance to accurately identify factors associated with the increased risk of progression and death, in order to develop effective follow-up and treatment strategies. However, to accurately assess the role of patients' specific characteristics in the progression of cancer several methodological challenges need to be overcome.

One difficulty, common to prognostic studies of cancer, concerns the need to separate the effects of prognostic factors on different clinical endpoints, such as disease recurrence vs recurrence-free death. Another difficulty, encountered in prognostic studies, is that the cause of death is not available or not accurately coded. Yet, some patients are likely to die of causes not related to the disease of primary interest, especially in cancers with longer survival and in those that affect older subjects. Until recently, the existing statistical methodology was not able to simultaneously, deal with both difficulties, i.e. to account for (i) possibly different effects of prognostic factors on death vs recurrence, and (ii) unknown causes of death. However, this challenge has been addressed by the recent development of the Markov relative survival model (MRS) , which extends the Markov multi-state model to incorporate relative survival modelling. Simulations demonstrate that MRS is able to accurately estimate different effects of prognostic factors on the risk of each of several events, including separate effects on disease-specific vs other causes of death. To date, the MRS had not been applied in clinical or epidemiological studies.

The aim of this study was to assess the potential advantages of the new multi-state relative survival model (MRS), proposed by Huszti et al. (2012), in a prognostic cancer study. To this end, we compared the MRS results with those obtained with two more conventional analyses, based on Cox's proportional hazards model, and the multi-state Markov model proposed by Alioum and Commenges (2001). The three models were applied to explore the impact of prognostic factors on cancer-specific mortality and recurrence, in a large population-based French registry of colorectal cancer, with up to 25 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

patient with primary digestive cancer between 1985 and 2000, TNM I-III, resected for cure, residing in Burgundy or Calvados, France

Exclusion Criteria:

metastatic cancer, non adenocarcinoma, recurrence within 6 month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with invasive colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 5194 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
death due to cancer | 10 years after resection
death due to recurrence | 10 years after resection

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France